CLINICAL TRIAL: NCT06519331
Title: M148 - Development of a New Method for Liver Stiffness Measurement Using FibroScan
Brief Title: Development of a New Method for Liver Stiffness Measurement Using FibroScan
Acronym: M148
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M148
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases
Keywords: FibroScan; Vibration Controlled Transient Elastography; Liver Stiffness Measurement
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patient (age >= 18 y.o) followed for a liver disease, all etiologies combined (Experimental): Adult patients followed in the Hepatology or Endocrinology department for a liver disease, suspected chronic liver disease or consequences of chronic liver disease, all etiologies combined.
  Interventions: Device: Research FibroScan (FS)

INTERVENTIONS:
Device: Research FibroScan (FS) — Patients #1 to #25:
  Exam 1: Examination with Research FibroScan. Exam 2: Examination with the Reference FibroScan at the same measurement point and with the same probe used for the Exam 1.
  Patients #26 to #75:
  Exam 1: Examination with the Research or Reference FibroScan. Exam 2: Examination with the Reference or Research FibroScan at the same measurement point and with the same probe used for the Exam 1.
  Patients #76 to #114:
  Exams 1 & 2: 2 consecutive examinations with the Research or Reference FibroScan.
  Exams 3 & 4: 2 consecutive examinations with the Reference or Research FibroScan at the same measurement point and with the same probe used for the Exams 1 & 2.

SUMMARY:
This is an European, prospective, interventional, multicenter clinical investigation that will take place in 2 French sites. 114 adults patients will be included. The study objective is to develop a new method for measuring liver stiffness using FibroScan.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) followed in the hepatology or endocrinology department for liver disease, suspected liver disease or consequences of liver disease, all etiologies combined.
* Adult patient able to give his written consent
* Patient affiliated to the French Social Security system

Exclusion Criteria:

* Vulnerable patients
* Patients with liver ascites
* Patients with heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Reduced intra-examination dispersion of liver stiffness measurements with the new measurement method. | 24 months

SECONDARY OUTCOMES:
Bias between the different stiffness measurements (reference/estimated reference/at rest) | 24 months
  Correlation coefficients will be done.
Bias between the estimated reference stiffness repetitions and between the stiffness at rest repetitions. | 24 months
  Intra-class correlation coefficients will be done.
Bias between the CAP measured with the Research FibroScan and the CAP measured with the Reference FibroScan | 24 months
  Correlation coefficients will be done.
Bias between the CAP repetitions done with the Research FibroScan | 24 months
  Intra-class correlation coefficients will be done.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupe Hospitalier Nord Essonne - Site Paris- Saclay, Orsay
  - Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region